CLINICAL TRIAL: NCT06585748
Title: The Effect of Lidocaine Spray Use on Patients Comfort in Undergoing Bladder Catheterization: a Prospective,observational ,controlled Study
Brief Title: Lidocaine Spray Use on Patients Comfort in Undergoing Bladder Catheterization
Status: Recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Elif Kaya Çelikel, MD, Ankara City Hospital Bilkent
Other Study IDs: ACH-Lidocaine
Record Dates: First submitted 2024-08-28; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Urinary Catheterization As the Cause of Abnormal Reaction of Patient, or of Later Complication, Without Mention of Misadventure At Time of Procedure
Keywords: Bladder catheterization; Pain control; Lidocaine spray; Patient comfort
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group L: Group L: Lidocaine spray. Lidocaine spray in our country is available in a 10% spray form, with each puff containing 10 mg of lidocaine. In Group L, 4 puffs of lidocaine spray were applied to the glans penis and urethral meatus, and after 5 minutes, the appropriate method and sterilization were used to apply a catheter gel, and a Foley catheter was placed in the bladder.
  Interventions: Drug: Lidocaine spray
- Group P: Group P: Placebo In Group P, 4 puffs of isotonic saline (%0.09 NaCl) spray were applied to the glans penis and urethral meatus, followed by catheter gel application and Foley catheter placement.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lidocaine spray — 4 puffs of lidocaine spray was applied to the glans penis and urethral meatus, and after 5 minutes, the appropriate method and sterilization were used to apply a catheter gel, and a Foley catheter was placed in the bladder. After bladder catheterization, pain scores were evaluated by a neutral emergency medicine physician at 0 minutes (during the procedure), and at 15, 30, and 60 minutes post-procedure. The Face Legs Arms Cry Consolability Pain Scale (FLACC) and Wong-Baker pain scales were used for this evaluation.
  Groups: Group L
Other: Placebo — No medication/application will be administered as placebo.
  Groups: Group P

SUMMARY:
Bladder catheterization is a procedure frequently performed in emergency departments and may cause symptoms such as pain and discomfort in patients. This study hypothesizes that lidocaine spray application will improve patient compliance and comfort from the outset and facilitate smoother medical procedures. In our prospective, case-controlled study, the patients were divided into two groups: Group L (lidocaine) and Group P (placebo). Pain conditions after bladder catheterization were evaluated at 0 minutes (during the procedure) and 15, 30 and 60 minutes after the procedure. Face Legs Arm Cry Consolability Pain Scale (FLACC) and Wong-Baker pain scales were used. All time periods in Group L, FLACC score and Wang Baker scores were found to be statistically significantly lower.The differences between the first measurement and the measurements at 15-30-60 minutes of the FLACC score were found to be significantly higher in group P than in group L. As a result, we recommend that lidocaine spray be applied before urinary catheter insertion. This study showed that lidocaine spray increased patients' sleep at the end and reduced the feeling of restlessness by reducing pain.

ELIGIBILITY:
Inclusion Criteria: The study included male patients over 18 years old, without trauma, with spontaneous urine output, and who were oriented and cooperative. -

Exclusion Criteria: Exclusion criteria were patients under 18 years old, female patients, patients with trauma, patients with globe vesicale (due to the need for rapid bladder catheterization), patients with anatomical variations, patients with urethral-bladder outlet problems preventing catheterization, and patients who refused to participate in the study.

-

Ages: 18 Years to 92 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of patients who required bladder catheterization during the follow-up and treatment process and came to the emergency departments of two major city hospitals in Ankara.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Lidocaine and Pain | 0., 15., 30., and 60. minutes
  The FLACC scale assesses acute pain based on facial expression, leg position, activity, crying, and consolability Each category is scored from 0-2, with 0 indicating a calm patient and 10 indicating a visibly distressed patient .

SECONDARY OUTCOMES:
Lidocaine and comfort | 0., 15., 30., and 60. minutes
  Wong-Baker pain scale evaluates pain based solely on facial expressions. A score of 0 represents no pain, while a score of 10 represents unbearable pain .

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No